CLINICAL TRIAL: NCT03438643
Title: Dynamic of Immunocompetent Populations in Patients Treated With Extracorporeal Photopheresis in Chronic Graft Versus Host Disease
Acronym: IMMUNO-PEC
Status: Terminated | Type: Observational
Why Stopped: lack of inclusions
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2017_29; 2017-A01889-44 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-01-29; First posted 2018-02-20 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Graft Versus Host Disease; Extracorporeal Photopheresis
Keywords: Graft versus host disease; Extracorporeal photopheresis; Immunomodulatory
MeSH Terms: conditions — Graft vs Host Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient: Patients treated with ECP and corticosteroid as first-line treatment for cGVHD
  Interventions: Diagnostic Test: Blood samples; Diagnostic Test: skin biopsy

INTERVENTIONS:
Diagnostic Test: Blood samples — Blood samples (42mL) will be taken before and during treatment.
Diagnostic Test: skin biopsy — skin biopsy will be taken before and during treatment.

SUMMARY:
Extracorporeal photopheresis (ECP) is a cellular therapy indicated in the treatment of chronic GVHD (cGVHD). In this study protocol, patients suffering from inaugural cGVHD will be treated with the association of ECP and corticosteroid treatment. Treatment will start by an induction stage with 2 sessions of ECP per week until the 10th week followed by a maintenance stage including one session every other week until the 22th week. The objective of this study is to highlight the immunological mechanism of extracorporeal photopheresis treatment. Indeed, ECP is based on an immunomodulatory immunological effect and despite several hypotheses highlighted by different teams; clear mechanisms still need to be defined. This French multicenter study realize an immunological follow-up before and during treatment to elucidate the impact of ECP on immune system of responder patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years who had a first allo-CSH for hematological pathology
* Body weight ≥ 40 kg.
* Confirmed diagnosis of inaugural cGVHD requiring systemic treatment.
* Any source of hematopoietic stem cells is allowed.
* All conditioning treatments are allowed.
* Patient validated by the local investigator as eligible for treatment with ECP according to the criteria of the investigating centers
* Patient treated according to the study plan with a ECP in 2 steps
* Patient having signed informed consent.
* Prophylaxis of GVH maintained during the onset of cGVHD is accepted.
* Effective contraception for men and women of childbearing age.

Exclusion Criteria:

* cGVHD ≥ 2nd line of treatment
* Exclusive pulmonary cGVHD
* cGVHD before J100
* cGVHD occurring after Donor Lymphocyte Injection (DLI)
* Overlaps syndrome aGVHD-cGVHD
* Late aGVHD
* Relapsed patient or progressive disease
* Non-controlled infection
* Second Allograft
* Leukopenia <0.5G / l at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with ECP and corticosteroid as first-line treatment for cGVHD.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2019-12-02 (Actual)

PRIMARY OUTCOMES:
Changes in circulating immunocompetent subsets for responder and non-responder patients treated with ECP in inaugural cGVHD. | at 6-week follow-up

SECONDARY OUTCOMES:
Changes in circulating immunocompetent subsets frequency for responder and non-responder patients treated with ECP in inaugural cGVHD. | at 22-week follow-up
Response rate (complete and partial response) according to NIH criteria | at 10 weeks and at 22 weeks
  Efficacy of ECP in inaugural cGVHD in combination with immunosuppressive therapy (prednisone + ciclosporin)
Comparison of serum and tissue biomarkers in responder and non-responder patients between the initial treatment and 6-week follow-up. | at baseline, at 6 week follow-up
QLQ-C30 version 3.0 | between 10-week and 22-week follow-ups.
  Evaluation of the quality of life for patients. QLQ-C30 is a composite score. QLQ-C30 Summary Score = (Physical Functioning+ Role Functioning+ Social Functioning+ Emotional Functioning+ Cognitive Functioning+ 10 0-Fatigue+ 100
  * Pain+ 100
  * Nausea_Vomiting+ 100
  * Dyspnoea+ 100
  * Sleeping Disturbances+ 100
  * Appetite Loss+ 100
  * Constipation+ 100
  * Diarrhoea)/13

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim YAKOU BAGHA, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Claude Huriez, CHU, Lille, France